CLINICAL TRIAL: NCT00816049
Title: Nordic Society of Paediatric Haematology and Oncology Treatment Protocol for Children (1.0 - 17.9 Years of Age) and Young Adults (18-45 Years of Age) With ALL. Efficacy of Individualised 6MP Dosing During Consolidation Therapy
Brief Title: ALL2008 Protocol for Childhood Acute Lymphoblastic Leukemia (ALL) - 6MP Consolidation Therapy
Acronym: ALL2008con
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Nordic Society for Pediatric Hematology and Oncology (Other)
Responsible Party: Principal Investigator, Kjeld Schmiegelow, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOPHO ALL2008 consolidation
Record Dates: First submitted 2008-12-23; First posted 2008-12-31 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: acute lymphoblastic leukemia; child; 6-mercaptopurine; minimal residual disease; efficacy; childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual | interventions — Mercaptopurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 6MPfixed (Active Comparator): Fixed dose 6-mercaptopurine days 30-85
  Interventions: Drug: 6MPfixed
- 6MPindividualized (Experimental): Individualized dose increments of 6-mercaptopurine days 30-85
  Interventions: Drug: 6MPindividualized

INTERVENTIONS:
Drug: 6MPindividualized — Oral 6-mercaptopurine with a starting dose of 25 mg/m2 and upward adjusted in steps of 25 mg/m2 (i.e. 50 or 75 mg/m2) if unacceptable bone-marrox toxicity is not encountered
  Other Names: PuriNethol, Puri-Nethol (6-mercaptopurine)
  Arms: 6MPindividualized
Drug: 6MPfixed — Oral 6-mercaptopurine at a fixed dose of 25 mg/m2 treatment days 30-85
  Other Names: PuriNethol, Puri-Nethol (6-mercaptopurine)
  Arms: 6MPfixed

SUMMARY:
The purpose of this study is to increase the fraction of patients, who become MRD-negative during consolidation for the non-HR ALL group through individualized intensification of the 6MP-dosage days 30-85.

DETAILED DESCRIPTION:
20% of children with ALL still fails to be cured. The ALL-2008 protocol is a treatment and research protocol that aims to improve the overall outcome of Nordic children and adolescents with ALL in comparison with the ALL-2000 protocol and previous NOPHO protocols.

The specific and primary objectives of the randomised study is:

To increase the fraction of patients, who become MRD-negative during consolidation for the non-HR ALL group through individualised intensification of the 6MP-dosage days 30-85. We will additionally measure EFS and toxicity as secondary end points of effect.

ELIGIBILITY:
Inclusion Criteria:

* Childhood ALL
* All mandatory biological data are available6
* Written informed consent has been obtained

Exclusion Criteria:

* Mixed lineage ALL
* Pre-treatment with glucocorticosteroids or other antileukemic agents for more than 1 week
* ALL predisposition syndromes
* Previous cancer
* Off protocol administration of additional chemotherapy during induction therapy
* Sexually active females not using contraception
* TPMT-deficiency

Ages: 1 Year to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 775 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2016-03-02 (Actual); Study Completion 2016-03-02 (Actual)

PRIMARY OUTCOMES:
Fraction of patients that become MRD-negative at treatment days 85 and/or 92 (end-of-consolidation) and event-free survival. MRD is measured either by Flow-cytometry (for PreB-ALL patients) or PCR for clonal generearrangements(for T-ALL patients) | 6 years

SECONDARY OUTCOMES:
Toxicity of treatment, degree of myelo-, hepato- and renal toxicity; and development of asparaginase antibodies. | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Schmiegelow, M.D., Study Chair — Rigshospitalet, Blegdamsvej 9, 2100 Copenhagen
Locations (6):
- Department of Pediatrics, Rigshospitalet, Copenhagen, Denmark
- Helsinki University Hospital, Helsinki, Finland
- University Hospital, Reykjavik, Iceland
- Trondheim University Hospital, Trondheim, Norway
- Sweden (2):
  - Department of Pediatrics, Drottning Sylvias Pediatric Hospital, Gothenburg
  - NOPHO nordic organisation for pediatric onology, Stockholm